CLINICAL TRIAL: NCT00652171
Title: Efficacy and Safety of Antidepressant Augmentation With Lamotrigine in Patients With Treatment-Resistant Depression
Brief Title: Efficacy and Safety of Antidepressant Augmentation With Lamotrigine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Social Security of the Civil Servants of Minas Gerais (Other Government)
Responsible Party: Milena Antunes Santos/Dr, Post - Graduation in Health Sciences, IPSEMG
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEP: 093/03
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Last update posted 2008-04-09 (Estimated); Status verified 2008-04

CONDITIONS: Depression
Keywords: Treatment; Augmentation; Resistant depression; Lamotrigine
MeSH Terms: conditions — Depression | interventions — Lamotrigine; Amides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 17 Patients - Mean age of 26 years old, 14 female and 3 male - with major depressive disorder in single or recurrent episodes, with moderate to severe intensity. Besides, They also had a history of treatment-resistant depression stage II or above according to the criteria of by Thase and Rush: failure to respond to treatment with at least 2 antidepressants of different classes, at the maximum tolerated dose for at least 6 weeks and absence of psychotic symptoms.
  Interventions: Drug: Lamotrigine
- 2 (Placebo Comparator): 17 Patients - 11 females and 6 males mean age of 29 years old - with major depressive disorder in single or recurrent episodes, with moderate to severe intensity. Besides, They also had a history of treatment-resistant depression stage II or above according to the criteria of by Thase and Rush: failure to respond to treatment with at least 2 antidepressants of different classes, at the maximum tolerated dose for at least 6 weeks and absence of psychotic symptoms.
  Interventions: Dietary Supplement: Amide

INTERVENTIONS:
Drug: Lamotrigine — Lamotrigine was added to the ongoing antidepressant. The doses were titrated to 200mg/day.
  Arms: 1
Dietary Supplement: Amide — Capsule of amide were given to this group of patients. They continued the ongoing antidepressants.
  Arms: 2

SUMMARY:
This study reports a clinical trial evaluating lamotrigine safety and efficacy as an antidepressant augmentation agent in treatment resistant depression, therefore adding more empirical evidence to the limited number of studies on the use of lamotrigine.

DETAILED DESCRIPTION:
Objective: This study reports a clinical trial evaluating lamotrigine safety and efficacy as an antidepressant augmentation agent in treatment resistant depression, therefore adding more empirical evidence to the limited number of studies on the use of lamotrigine.

Method: A double-blind pilot study was conducted with 34 nonbipolar, nonpsychotic patients who had DSM-IV major depressive disorder and were resistant to at least 2 antidepressants. The subjects were on taking antidepressant therapy and were randomly assigned to receive placebo or lamotrigine as an adjunct therapy for 8 weeks. They were evaluated on a biweekly basis in order to access assess the efficacy and the safety of the drug.

ELIGIBILITY:
Inclusion Criteria:

* They were selected according to a clinical interview based on DSM-IV criteria for major depressive disorder in single or recurrent episodes, with moderate to severe intensity. Besides
* They also had a history of treatment-resistant depression stage II or above according to the criteria of by Thase and Rush11

  * failure to respond to treatment with at least 2 antidepressants of different classes
  * at the maximum tolerated dose for at least 6 weeks and absence of psychotic symptoms

Exclusion Criteria:

* Pregnant or lactating women or those capable of getting pregnant that who were not using contraceptive methods were excluded as well as patients with severe clinical diseases or organic mental disorder
* Further exclusion criteria were acute depression with risk of suicide
* psychosis
* and bipolar disorder as well as personality disorders and disorders related to alcohol and other drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2004-01; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Montgomery and Asberg Scale for Depression | 8 weeks

SECONDARY OUTCOMES:
Clinical Global Impression | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Milena A Santos, Master, Principal Investigator — City Hall of Beló Horizonte; Claudia Hara, Master, Study Chair — Faculdade de Saúde e Ecologia Humana; Fabio L Rocha, PhD, Study Director — Institute of Social Security of the Civil Servants of Minas Gerais

REFERENCES:
- [Background] Barbosa L, Berk M, Vorster M. A double-blind, randomized, placebo-controlled trial of augmentation with lamotrigine or placebo in patients concomitantly treated with fluoxetine for resistant major depressive episodes. J Clin Psychiatry. 2003 Apr;64(4):403-7. doi: 10.4088/jcp.v64n0407. PMID 12716240
- [Background] Rocha FL, Hara C. Lamotrigine augmentation in unipolar depression. Int Clin Psychopharmacol. 2003 Mar;18(2):97-9. doi: 10.1097/00004850-200303000-00006. PMID 12598821
- [Background] Barbee JG, Jamhour NJ. Lamotrigine as an augmentation agent in treatment-resistant depression. J Clin Psychiatry. 2002 Aug;63(8):737-41. doi: 10.4088/jcp.v63n0813. PMID 12197456
- [Derived] Santos MA, Rocha FL, Hara C. Efficacy and safety of antidepressant augmentation with lamotrigine in patients with treatment-resistant depression: a randomized, placebo-controlled, double-blind study. Prim Care Companion J Clin Psychiatry. 2008;10(3):187-90. doi: 10.4088/pcc.v10n0302. PMID 18615166
- See also: FDA, Overview of Lamotrigine — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm?fuseaction=Search.Overview&DrugName=LAMOTRIGINE